CLINICAL TRIAL: NCT03298841
Title: Zeiss Lumera Microscope With Callisto Software
Brief Title: Clinical Comparison of Length of Cataract Procedures With Zeiss Lumera Versus Older Zeiss Microscope
Status: Completed | Type: Observational
Sponsor: Toyos Clinic (Other)
Responsible Party: Principal Investigator, Melissa Toyos, Principal Investigator, Toyos Clinic
Other Study IDs: ZEISS-2017-003
Record Dates: First submitted 2017-09-22; First posted 2017-10-02 (Actual); Results first posted 2021-04-22 (Actual); Last update posted 2021-04-22 (Actual); Status verified 2021-04

CONDITIONS: Cataract
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Zeiss — This study proposal will highlight the advanced technology features of the Zeiss Lumera surgical operating microscope which include but are not limited to:
  Stereo Coaxial Illumination for improved visualization High resolution video screen/co-observation tool to help OR staff anticipate next steps Integrated toric alignment tool Surgical microscope touch screen Cordless foot control for faster turnover between cases

SUMMARY:
Study design will be a mix of retrospective (older Zeiss microscope previously in use at our surgery center) and prospective data collection with the Lumera and Callisto software.

The Lumera and Callisto software system will be used for all cataract surgeries including toric analyses and lens placement.

DETAILED DESCRIPTION:
Needs Assessment

Research on this topic is needed as over 3 million cataract surgeries are performed in the United States each year. The number of surgeries performed is growing as baby boomers age. Reimbursements continue to decline, necessitating ever improving operating and surgical efficiencies in the operating room setting for physicians and small business owners to remain financially viable. New governmental regulations dictate that physician payments will be related to patient satisfaction and outcomes which may be better provided by newer and better surgical technologies.

The Lumera operating microscope and Callisto software system provide several features that may enhance operating room flow including HD video screen and co-observant microscopes that can be independently adjusted to help operating room staff anticipate the needs of the surgeon. Enhanced retroillumination would be expected to translate into fewer complications and more confidence during surgery which could lead to less operating time, phaco energy used and improved visual outcomes. The toric alignment assistance device may lead to more accurate toric placement and improved visual outcomes after surgery.

Target audience would include all cataract surgeons both high and lower volume.

There is currently a dearth of published literature on this technology and its benefits in routine cataract surgery. There are no registered similar trials on Clinicaltrials.gov

ELIGIBILITY:
Inclusion Criteria:

* Visually significant cataract

Exclusion Criteria:

* Not visually significant cataract

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 patients with visually significant cataracts
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2017-09-20 (Actual); Study Completion 2017-09-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Toyos, md, Principal Investigator — Toyos Clinic
Locations (1):
- Toyos Clinic, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Zeiss Group: patients undergoing uncomplicated phacoemulsification using Zeiss Lumera microscope with Callisto software
- Leica Stativ S3B: patients undergoing uncomplicated phacoemulsification using Leica Stativ S3B microscope
Period: Overall Study
Arm/Group | Zeiss Group | Leica Stativ S3B
Started | 25 | 25
Completed | 25 | 25
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: sequential series of patients with uncomplicated cataracts undergoing phacoemulsification at one surgery site
Groups:
- Total: Total of all reporting groups
Arm/Group | Zeiss Group | Leica Stativ S3B | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 23 | 45
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 16 | 31
  Male | 10 | 9 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Improvement in Operating Room Efficiencies During Cataract Surgery With the Use of the New Lumera Operating Microscope Versus an Older Zeiss Model Operating Scope
Description: operating times during cataract surgery will be measured with the use of the new Lumera operating microscope versus an older Zeiss model operating scope by two experienced cataract surgeons in a single surgery center
Time Frame: during surgery assessed up to one hour
Population: patients undergoing uncomplicated phacoemulsification by two surgeons at one surgery site
Measure: Mean (Standard Deviation); unit: minutes per surgical procedure
Arm/Group | Zeiss Group | Leica Stativ S3B
Number analyzed (Participants) | 25 | 25
minutes per surgical procedure | 11.15 (2.42) | 14.18 (8.67)

2. Secondary Outcome: Number of Serious Adverse Events During Intra-operative and Post-operative Period
Description: events that are life or vision threatening, that require hospitalization or permanent disability of any type
Time Frame: 6 weeks
Population: patients scheduled for routine cataract surgery with one of two experienced surgeons
Measure: Count of Participants; unit: Participants
Groups:
- Cataract Surgery Patients: Patients undergoing immediate cataract surgery at a single site with one of two operating microscopes
Arm/Group | Cataract Surgery Patients
Number analyzed (Participants) | 50
Participants | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Zeiss Group | Leica Stativ S3B
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25
Other Adverse Events (participants affected / at risk) | 0/25 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: and Statistical Analysis Plan (2017-09-22): https://cdn.clinicaltrials.gov/large-docs/41/NCT03298841/Prot_001.pdf
  • Statistical Analysis Plan (2020-12-09): https://cdn.clinicaltrials.gov/large-docs/41/NCT03298841/SAP_002.pdf
  • Informed Consent Form (2017-01-20): https://cdn.clinicaltrials.gov/large-docs/41/NCT03298841/ICF_003.pdf